CLINICAL TRIAL: NCT03239327
Title: Vaginal Misoprostol Before Elective Cesarean Section to Improve Neonatal Respiratory Outcomes . Randomized Controlled Clinical Study
Brief Title: Vaginal Misoprostol to Improve the Neonatal Respiratory Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Makhlouf, Professor.Ahmed Mohammed Ahmed Makhlouf, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: assiut university women health
Record Dates: First submitted 2017-07-30; First posted 2017-08-04 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-08

CONDITIONS: Neonatal Respiratory Distress
Keywords: Misoprostol; neonatal; respiratory distress; cesarean section
MeSH Terms: conditions — Pulmonary Atelectasis; Dyspnea | interventions — Misoprostol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): For the study group the enrolled women will receive 50 microgram misoprostol vaginally 60 minutes before CS
  Interventions: Drug: Misoprostol
- control group (No Intervention): For the control group mothers enrolled will receive nothing.

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Prostaglandin E1,Cytotec
  Arms: study group

SUMMARY:
Project summary:

Objective: To test the hypothesis that administration of vaginal Misoprostol before elective cesarean section will improve the neonatal respiratory outcomes in late preterm and early term neonates through induction of catecholamine surge.

Design: Randomized controlled clinical trial. Setting: Women health center ,Assiut university hospital. Patients: mothers planned for cesarean section at 34 - 37weeks. Intervention: two hundred and ninety two women will be randomly allocated to receive either 50 micrograms of Misoprostol per vagina within one hour before cesarean section (study group; n= 146) or receive nothing (control group; n = 146) .

Main outcome measure: Apgar score at 1 and 5 minutes.

DETAILED DESCRIPTION:
Methodology: After a written informed consent obtained, women who are fitting the inclusion criteria will be randomly allocated using sealed, coded, opaque and sequentially numbered envelopes containing computer generated random numbers into either the study group or the control group. For the study group the enrolled women will receive 50 microgram misoprostol vaginally within 60 minutes before CS. For the control group mothers enrolled will receive nothing.

Observation and data collection: Cardiotocographic monitoring will be undertaken after maternal misoprostol administration to detect any evidence of uterine hyperstimulation and fetal distress.

Ritodrine IV will be used as a tocolytic agent in case of uterine tachysystole. 100 mg of ritodrine will be added to 500 ml of 0.5% dextrose, the solution will be administered as following:

5 drops / minute in the 1st 10 minutes. 10 drops / minute in the next 10 minutes then 15 drops / minute . The clinician should adjust the infusion rate so that the pulse rate doesn't exceed 120b/min and lung bases are free of crepitations.

The surgical and anesthetic teams will be in a state of complete readiness for the ECS from the time of maternal misoprostol administration after enrollment. Details on maternal fluid-electrolyte status during ECS will be recorded as maternal fluid overload is reported to be associated with respiratory distress in the newborn. (SinghiS,Chookang E;1984) blood loss during and 1 hour after the operation will be estimated.

Maternal data: Patient name, hospital number, age, parity, gestational age, any medical disorder and indication of CS.

Neonatal observations: delivery room care details will be noted, neonatal heart rate, respiratory rate, and signs of respiratory distress- for example, grunting, chest wall retractions, nasal flaring- will be recorded hourly in the postnatal ward for eight hours and once only at 24 hours of age after delivery. Management of a neonate with respiratory distress (defined as respiratory rate at rest.60/min and/or signs of respiratory distress) will be left to the neonatal team. Severity of illness, provisional and final diagnosis, and outcome (death/discharge home/transfer to other hospital) will be recorded if any neonate would be admitted to the neonatal intensive care unit for respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

All pregnant women who are planned for elective (planned& pre labor) cesarean section at 34 -37 weeks gestation.

Exclusion Criteria:

1. Pregnancies with known fetal malformation/s or chromosomal aberrations.
2. Presence of absolute contraindication for use of misoprostol.(i.e known hypersensitivity to the drug)
3. Women before 34 and after 37 weeks gestation .
4. Non reassuring cardiotocogram immediately before recruitment.
5. multiple pregnancies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
1- Rate of Neonatal Intensive Care Unit admission for neonatal respiratory distress. | During the first 24 hours of life.
  The number of neonates who need Neonatal Intensive Care Unit admission in each study group

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Makhlouf, professor, Principal Investigator — women health center,Assiut university,Assiut,Egypt
Locations (1):
- women health center,Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Motaze NV, Mbuagbaw L, Young T. Prostaglandins before caesarean section for preventing neonatal respiratory distress. Cochrane Database Syst Rev. 2013 Nov 11;2013(11):CD010087. doi: 10.1002/14651858.CD010087.pub2. PMID 24218013
- [Background] Singh M, Patole S, Rane A, Naidoo D, Buettner P. Maternal intravaginal prostaglandin E2 gel before elective caesarean section at term to induce catecholamine surge in cord blood: randomised, placebo controlled study. Arch Dis Child Fetal Neonatal Ed. 2004 Mar;89(2):F131-5. doi: 10.1136/adc.2002.025957. PMID 14977896
- [Background] Hansen AK, Wisborg K, Uldbjerg N, Henriksen TB. Risk of respiratory morbidity in term infants delivered by elective caesarean section: cohort study. BMJ. 2008 Jan 12;336(7635):85-7. doi: 10.1136/bmj.39405.539282.BE. Epub 2007 Dec 11. PMID 18077440
- [Background] Yang JY, Fang LJ, Tsou Yau KI. Labor pain before elective cesarean section reduces neonatal respiratory distress. Zhonghua Min Guo Xiao Er Ke Yi Xue Hui Za Zhi. 1997 Jan-Feb;38(1):38-43. PMID 9066188